CLINICAL TRIAL: NCT07322081
Title: Effect of a Mindfulness-Based Stress Reduction Program for Caregivers of Individuals With Chronic Mental Illness on Cognitive Control and Flexibility , Psychological Well-Being and Self-Compassion
Brief Title: Effect of a Mindfulness-Based Stress Reduction Program on Caregivers
Acronym: MBSR-CG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ömer USLU, PhD Student in Psychiatric Nursing, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MBSR-Caregivers-2025; PhD-Thesis-2025 (Other: Aydın Adnan Menderes University)
Record Dates: First submitted 2025-07-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Caregiver Stress in Chronic Mental Illness; Psychosocial Burden in Psychiatric Caregivers; Chronic Mental Illness Caregiving; Cognitive and Emotional Outcomes in Caregivers; Mental Illness Caregiver Support
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial with a parallel assignment model. Eligible participants are planned to be randomly assigned to either an intervention group receiving the Mindfulness-Based Stress Reduction program or a control group receiving usual care throughout the study period.
Masking Description: Due to the nature of the behavioral intervention, masking of participants and care providers is not feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction Program (Experimental): Participants assigned to this arm receive the Mindfulness-Based Stress Reduction (MBSR) program designed for primary caregivers of individuals with chronic mental illnesses, in addition to routine services provided by the community mental health center.
  Interventions: Behavioral: The Mindfulness-Based Stress Reduction program consists of structured mindfulness practices, psychoeducation, and experiential exercises delivered to caregivers.; Other: Usual Care Group
- Control Group (Usual Care) (No Intervention): Participants assigned to this arm receive routine care and standard support services provided by the community mental health center and do not receive the Mindfulness-Based Stress Reduction program.

INTERVENTIONS:
Behavioral: The Mindfulness-Based Stress Reduction program consists of structured mindfulness practices, psychoeducation, and experiential exercises delivered to caregivers. — The Mindfulness-Based Stress Reduction (MBSR) program is a structured behavioral intervention designed for primary caregivers of individuals with chronic mental illnesses. The program includes mindfulness practices, psychoeducation, and experiential exercises aimed at increasing present-moment awareness and adaptive coping skills. Sessions are delivered in a group format according to a standardized program structure.
  Arms: Mindfulness-Based Stress Reduction Program
Other: Usual Care Group — Usual care consists of standard support and services routinely provided by the community mental health center.
  Other Names: Standard Care
  Arms: Mindfulness-Based Stress Reduction Program

SUMMARY:
This study is designed to investigate the effects of a Mindfulness-Based Stress Reduction (MBSR) program on cognitive control and flexibility, psychological well-being, and self-compassion among primary caregivers of individuals with chronic mental illnesses. Caregivers of individuals with chronic mental health conditions are exposed to prolonged psychological, emotional, and cognitive demands, which may negatively affect their mental well-being and coping capacities.

The study adopts a mixed-methods approach using an exploratory sequential design in order to obtain a comprehensive understanding of caregivers' needs and experiences and to evaluate the potential impact of the intervention. Qualitative findings are intended to inform the development and structuring of the MBSR program, while the quantitative phase is designed to examine changes in key psychological outcomes following the intervention. The study aims to contribute to the growing body of evidence supporting mindfulness-based interventions for caregiver populations and to inform future mental health service practices.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effects of a Mindfulness-Based Stress Reduction (MBSR) program on cognitive control and flexibility, psychological well-being, and self-compassion in primary caregivers of individuals with chronic mental illnesses receiving services from a community mental health center. Caregiving for individuals with chronic mental health conditions often involves sustained emotional, cognitive, and social demands, which may increase vulnerability to psychological distress and reduce adaptive coping capacities.

The study is designed as a mixed-methods research utilizing an exploratory sequential design, integrating qualitative and quantitative research components. In the initial qualitative phase, in-depth, face-to-face interviews are planned to explore caregivers' experiences, perceived challenges, coping strategies, and expectations related to caregiving and psychological support. The qualitative findings are intended to guide the development, adaptation, and content refinement of the MBSR intervention in accordance with the specific needs of the caregiver population.

Following the qualitative phase, the quantitative component of the study is designed as a randomized controlled experimental trial. Eligible caregivers are planned to be randomly assigned to either an intervention group receiving the MBSR program or a control group receiving routine services. The MBSR program is structured to include mindfulness practices, psychoeducation, and experiential exercises aimed at enhancing present-moment awareness, emotional regulation, cognitive flexibility, and self-compassion.

Standardized self-report instruments are planned to be used to assess cognitive control and flexibility, psychological well-being, and self-compassion at predefined assessment points. The quantitative findings are intended to complement the qualitative results and to provide a systematic evaluation of the potential effects of the MBSR program.

The integration of qualitative and quantitative findings is expected to provide a comprehensive understanding of the intervention process and outcomes, supporting the development of evidence-based psychosocial interventions for caregivers of individuals with chronic mental illnesses within community mental health service settings.

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregiver of an individual with a chronic mental illness who is registered at the Community Mental Health Center (CMHC) of Söke Fehime Faik Kocagöz State Hospital
* Residing in the Söke district of Aydın province
* Being literate
* Having been the primary caregiver of the patient for at least six months

Exclusion Criteria:

* Having been diagnosed with any psychiatric disorder
* Having an intellectual disability
* Data from caregivers who submitted incomplete data collection forms were excluded from the study
* Caregivers who chose to withdraw from the study during the research process were excluded, and any data obtained from them were not used in the analysis
* Individuals who missed more than two sessions of the Mindfulness-Based Stress Reduction Program were excluded, and their data were not included in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Cognitive Control and Flexibility Questionnaire (CCFQ) | Baseline, immediately post-intervention, and 3-month follow-up
  Cognitive Control and Flexibility (Cognitive Control and Flexibility Questionnaire) Outcome Measure Description: Cognitive control and flexibility are assessed using the Cognitive Control and Flexibility Questionnaire (CCFQ), a self-report scale designed to evaluate caregivers' perceived ability to regulate thoughts and behaviors and to adapt flexibly to changing environmental demands. The total score ranges from 18 to 126, with higher scores indicating greater cognitive control and flexibility.

SECONDARY OUTCOMES:
Psychological Well-Being Scale (PWBS) | Baseline, immediately post-intervention, and 3-month follow-up
  Psychological well-being is assessed using the Psychological Well-Being Scale (PWB Scale), a self-report instrument that measures multiple dimensions of well-being, including autonomy, personal growth, purpose in life, self-acceptance, environmental mastery, and positive relations with others. The scale consists of 42 items rated on a 6-point Likert scale, yielding a total score ranging from 42 to 252, with higher scores indicating greater psychological well-being.

OTHER OUTCOMES:
Self-Compassion Scale - Short Form (SCS-SF) | Baseline, immediately post-intervention, and 3-month follow-up
  Self-compassion is assessed using the Self-Compassion Scale-Short Form (SCS-SF), a self-report instrument designed to measure individuals' self-kindness, common humanity, and mindfulness in response to personal difficulties. The scale consists of 12 items rated on a 5-point Likert scale, yielding a total score ranging from 12 to 60, with higher scores indicating greater levels of self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Söke Fehime Faik Kocagöz State Hospital Community Mental Health Center, Aydin, Söke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The anonymized individual participant data (IPD) that underlie the results reported in this study, including demographic characteristics, outcome measures, and group assignment, will be shared with qualified researchers upon reasonable request. Personal identifiers will be removed to ensure confidentiality and compliance with ethical standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the study results and will remain accessible for a period of 5 years. Researchers interested in accessing the data must submit a formal request and sign a data use agreement.
Access Criteria: Access to the anonymized IPD and supporting documents will be granted to academic researchers or institutions conducting non-commercial scientific studies. Requests should be made in writing to the corresponding author and must include a research proposal. Approved users will be required to sign a data-sharing agreement ensuring confidentiality and appropriate data use.

REFERENCES:
- See also: No external links are available at this time. — https://www.adu.edu.tr
- Available data/document: Study Protocol — https://www.adu.edu.tr — No external links to the study data are publicly available at this time. Data requests can be made by contacting the corresponding author or the Community Mental Health Center at Aydın Adnan Menderes University.